CLINICAL TRIAL: NCT00001193
Title: A Multimodality Treatment Approach to Patients With Inflammatory Cancer of the Breast and Locally Advanced Non-Inflammatory Stage III Breast Cancer and Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 840216; 84-C-0216
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-08

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
Keywords: Autologous; Melphalan; Stage III; Transplantation
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Melphalan

INTERVENTIONS:
Procedure: high dose melphalan and autologous bone marrow transplantation

SUMMARY:
This study is designed to evaluate the efficacy of high dose melphalan and autologous bone marrow transplantation given as consolidation therapy to patients with inflammatory or metastatic carcinoma of the breast in complete remission. All patients entered will receive induction therapy with cyclophosphamide, adriamycin, methotrexate and 5-fluorouracil with hormonal synchronization utilizing tamoxifen and premarin as in a previous Medicine Branch protocol (MB-160C). Among patients with inflammatory carcinoma of the breast, pathologic complete responders will receive irradiation to the breast and regional lymph nodes; convertible partial responders and clinical complete responders with residual disease on biopsy will undergo surgical resection of bulk disease followed by irradiation of the chest wall and regional lymph nodes excluding the axilla. Both groups of responders will be randomized to receive either systemic consolidation therapy with high dose melphalan (180 mg/M2 total dose over 3 days) and autologous bone marrow transplantation followed by maintenance therapy or maintenance therapy alone. Complete responders in this noninflammatory group will not receive further therapy since, historically, they have done well following induction and local therapy, with maintenance therapy alone.

Patients with metastatic breast cancer will be assessed for response throughout induction therapy. Complete and convertable partial responders will receive consolidative therapy and be randomized to ABMT followed by 6 months of maintenance therapy vs. maintenance alone.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy of high dose melphalan and autologous bone marrow transplantation given as consolidation therapy to patients with inflammatory or metastatic carcinoma of the breast in complete remission. All patients entered will receive induction therapy with cyclophosphamide, adriamycin, methotrexate and 5-fluorouracil with hormonal synchronization utilizing tamoxifen and premarin as in a previous Medicine Branch protocol (MB-160C). Among patients with inflammatory carcinoma of the breast, pathologic complete responders will receive irradiation to the breast and regional lymph nodes; convertible partial responders and clinical complete responders with residual disease on biopsy will undergo surgical resection of bulk disease followed by irradiation of the chest wall and regional lymph nodes excluding the axilla. Both groups of responders will be randomized to receive either systemic consolidation therapy with high dose melphalan (180 mg/M2 total dose over 3 days) and autologous bone marrow transplantation followed by maintenance therapy or maintenance therapy alone. Complete responders in this noninflammatory group will not receive further therapy since, historically, they have done well following induction and local therapy, with maintenance therapy alone.

Patients with metastatic breast cancer will be assessed for response throughout induction therapy. Complete and convertable partial responders will receive consolidative therapy and be randomized to ABMT followed by 6 months of maintenance therapy vs. maintenance alone.

ELIGIBILITY:
Patients must have a histologically documented diagnosis of mammary carcinoma and evaluable disease in the breast.

Diagnostic tissue must be reviewed at NIH.

All ICB patients must meet Haagensen's clinical criteria of ICB.

Patients with metastatic breast cancer must have evaluable disease.

There must be no history of prior cytotoxic therapy.

There must be no history of previous malignancy except for cured nonmelanoma skin cancer and cervical carcinoma in situ.

Performance status (Karnofsky scale) must be greater than 30 for patients with metastatic breast cancer.

Staging workup must be negative for distant metastases in Stage III patients.

WBC count greater than 4000 per mm(3) and platelet count greater than 100,000 per mm(3).

Normal hepatic and renal function, unless due to tumor involvement.

Patients must be willing to give informed consent and be geographically accessible for follow up.

No history of other malignant neoplasms except for curatively treated nonmelanoma skin cancer or surgically cured carcinoma of the cervix in situ.

Patients must not be poor medical or psychiatric risks because of non-malignant systemic disease which would preclude them being subjected to any of the treatments in this protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 1984-11; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Chu AM, Wood WC, Doucette JA. Inflammatory breast carcinoma treated by radical radiotherapy. Cancer. 1980 Jun 1;45(11):2730-7. doi: 10.1002/1097-0142(19800601)45:113.0.co;2-c. PMID 6769583
- [Background] Buzdar AU, Montague ED, Barker JL, Hortobagyi GN, Blumenschein GR. Management of inflammatory carcinoma of breast with combined modality approach - an update. Cancer. 1981 Jun 1;47(11):2537-42. doi: 10.1002/1097-0142(19810601)47:113.0.co;2-x. PMID 6790155
- [Background] McElwain TJ, Hedley DW, Gordon MY, Jarman M, Millar JL, Pritchard J. High dose melphalan and non-cryopreserved autologous bone marrow treatment of malignant melanoma and neuroblastoma. Exp Hematol. 1979;7 Suppl 5:360-71. PMID 400698